CLINICAL TRIAL: NCT05509036
Title: Frailty, Outcomes, Recovery and Care Steps of Critically Ill Patients (FORECAST) Multi-Center Study
Brief Title: Frailty, Outcomes, Recovery and Care Steps of Critically Ill Patients (FORECAST) Study Multi-Center Study
Acronym: FORECAST
Status: Completed | Type: Observational
Sponsor: Dr. John Muscedere (Other)
Collaborators: Canadian Frailty Network (Other)
Responsible Party: Sponsor-Investigator, Dr. John Muscedere, Professor of Medicine, Queen's University
Organization: Queen's University (Other)
Other Study IDs: FORECAST, V4 - June 7, 2019
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-09

CONDITIONS: Frailty; Critical Illness
Keywords: Outcomes; Frailty
MeSH Terms: conditions — Frailty; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Critically ill adults > 50 admitted to the ICU and receiving a life support intervention
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
A prospective observational study of critically ill patients over the age of 50, studying the occurrence of frailty as measured by a variety of frailty measures, processes of care and long term outcomes.

DETAILED DESCRIPTION:
Frailty is common in critically ill elderly patients, and is associated with adverse impacts on outcomes and is becoming increasingly common in Intensive Care Unit (ICU) populations. However it is not clear as to how to best measure frailty and when to do so. It is also not clear as to how processes of care impact on the outcomes observed. We hypothesize that frailty in survivors of critical illness will be measurable at hospital discharge, will correlate with processes of care while in ICU and will better discriminate long term outcomes when compared to severity of illness or the degree of frailty present on ICU admission.

ELIGIBILITY:
Inclusion Criteria:

Must Meet both 1 and 2

* 1. Age > 50 years. We have selected >50 years in keeping with prior descriptions of critically ill patients [17].

  2. Receipt of at least one of the following life support interventions for over 24 hours:
  1. Mechanical ventilation: Both invasive and non-invasive either solely or in combination are acceptable. High flow oxygen (e.g. OPTIFLOW) as a form of Non-Invasive Ventilation (NIV) is acceptable but the patient's Fraction of Inspired Oxygen (FIO2) at the time of enrollment must be greater > 50%.
  2. Vasoactive medications (vasopressors or inotropes).
  3. Acute renal replacement therapy (RRT). Patient must have been admitted to ICU for the receipt of renal replacement therapy, either intermittent or continuous and after 24 hours of ICU admission, there is a continued need for further RRT.

Exclusion Criteria:

1. ICU admission greater than 5 days at the time of enrollment.
2. Expected to survive for less than 72 hours after study enrollment.
3. No family or caregivers available to collect collateral history.
4. Family or caregivers not able to speak English or French.
5. Projected inability to complete 6 month follow-up either by telephone or in-person.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients over the age of 50 receiving life support interventions in the Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Frailty status | 6 Months
  Frailty as measured with the Clinical Frailty Scale (CFS). CFS is a 9 point scale with frailty defined as a CFS > 4 with higher scores indicating greater degrees of frailty.
Frailty status | 6 Months
  Frailty as measured with the Frailty Index (FI). The FI is indicated by the proportion of deficits present over the number measured and is scored as a fraction between 0 and 1.0. Frailty is considered to be present when the FI is > 0.20 and the severity of frailty is considered higher with increasing values for the FI.

SECONDARY OUTCOMES:
Number of patients with a measure of frailty prior to hospital discharge. | 28 days
  Measure of the Frailty Index and Clinical Frailty Scale prior to discharge
Correlation of frailty severity at hospital discharge with long term outcomes (mortality, Quality of Life and Need for Institutionalization) | 6 months
  Clinical outcomes at 6 months will include mortality, Quality of Life (EQ5L) and need for Institutionalization
Impact of admission critical illness on the development and severity of frailty as measured by a Frailty Index or Clinical Frailty Scale | 28 days and 6 months
  Correlation with the progression or presence of frailty as measured with the Frailty Index or Clinical Frailty Scale
Correlation of ICU processes of care (nutritional adequacy, adverse events, mobilization and sedation) with frailty progression as measured by the Clinical Frailty Scale or Frailty Index | 28 days
  Correlation of processes of care in ICU with frailty progression

CONTACTS AND LOCATIONS:
Overall Officials: John Muscedere, MD, Principal Investigator — Queens University
Locations (11):
- Canada (11):
  - University of Alberta, Edmonton, Alberta
  - Dalhousie University - QEII, Halifax, Ontario
  - St Joe's Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Center, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Laval University, Laval, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Maisonneuve Rosemont, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No